CLINICAL TRIAL: NCT03813992
Title: A Phase III, Dose Ranging, Multi-centre, Randomised, Double Blind, Placebo Controlled, Home Use, Parallel Group Clinical Trial of Topically-applied Glyceryl Trinitrate for the Treatment of Erectile Dysfunction, With an Open Label Extension
Brief Title: Clinical Trial Using Topically Applied Glyceryl Trinitrate (GTN) for the Treatment of Erectile Dysfunction
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Futura Medical Developments Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FM57
Record Dates: First submitted 2019-01-15; First posted 2019-01-23 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2022-02

CONDITIONS: Erectile Dysfunction
MeSH Terms: conditions — Erectile Dysfunction | interventions — Nitroglycerin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- MED2005 0.2% (Active Comparator): MED2005 0.2% w/w gel to deliver 0.6 mg dose of GTN applied topically prior to a sexual intercourse attempt
  Interventions: Drug: MED2005
- MED2005 0.4% (Active Comparator): MED2005 0.4% w/w gel to deliver 1.2 mg dose of GTN applied topically prior to a sexual intercourse attempt
  Interventions: Drug: MED2005
- MED2005 0.6% (Active Comparator): MED2005 0.6% w/w gel to deliver 1.8 mg dose of GTN applied topically prior to a sexual intercourse attempt
  Interventions: Drug: MED2005
- Placebo vehicle (Placebo Comparator): Placebo vehicle applied topically prior to a sexual intercourse attempt
  Interventions: Drug: MED2005

INTERVENTIONS:
Drug: MED2005 — Topical Product
  Other Names: Glyceryl Trinitrate

SUMMARY:
To demonstrate the efficacy of various doses of MED2005 versus placebo in male patients with clinically diagnosed erectile dysfunction, and to evaluate the long-term efficacy and safety (12 months) of MED2005.

DETAILED DESCRIPTION:
A phase III, dose-ranging, multi-centre, randomised, double-blind, placebo controlled , home-use, parallel group clinical trial of topically applied glyceryl trinitrate for the treatment of erectile dysfunction with an open label extension

ELIGIBILITY:
Inclusion Criteria:

1. Subject is a male aged between 18 and 70 years inclusive, at screening
2. Confirmed clinical diagnosis of ED for more than 3 months according to the NIH Consensus Statement ('the inability to achieve or maintain penile erection sufficient for satisfactory sexual performance at least once')
3. Subject answers 'yes' to the question regarding the presence of residual EF over the past 3 months: 'At home over the past 3 months, have you experienced at least some growth of your penis in response to: (1) mechanical stimulation by yourself or your partner, or (2) visual stimulation?'
4. Subject has been involved in a continuous heterosexual relationship for at least 6 months prior to screening
5. Documented written informed consent from both subject and his female partner
6. If the male subject's female partner is of childbearing potential from the time of first sexual intercourse attempt during the screening period until the last administration of study treatment, then the couple must have been using a medically acceptable form of contraception for at least 3 months prior to entering the study, and agree to continue such use for at least 1 month after the last study drug administration. Subjects who are or wish to become pregnant will not be included in the study.
7. Subject and his female partner are capable of understanding and complying with the requirements of the protocol and must have signed the ICF prior to participation in any study related procedures
8. Low IIEF-EF scores (≤ 25) during the screening period

To continue in the open-label extension phase of the study, subjects must meet the following inclusion criteria at the follow-up visit of the double-blind phase (Visit 6):

1. Subject and his female partner complete the double-blind phase
2. Subject and his female partner were compliant to study procedures during the double blind phase
3. Documented written informed consent from both subject and his female partner
4. If the male subject's female partner is of childbearing potential from the time of first sexual intercourse attempt during the screening period until the last administration of study treatment, then the couple must have been using a medically acceptable form of contraception for at least 3 months prior to entering the study, and agree to continue such use for at least 1 month after the last study drug administration. Subjects who are or wish to become pregnant will not be included in the study.

Exclusion Criteria:

1. Any significant or serious cardiovascular, pulmonary, hepatic, renal, gastrointestinal, haematological, endocrinological, metabolic, neurological or psychiatric disease which, in the opinion of the PI, renders the subject unfit to take part in the study
2. Subject has any history of an unstable medical or psychiatric condition or using any medication that, in the opinion of the PI, is likely to affect the subject's ability to complete the study or precludes the subject's participation in the study Certain concomitant medications; e.g. other vasodilators, calcium channel blockers, angiotensin converting enzyme (ACE) inhibitors, beta blockers, diuretics, anti hypertensives, tricyclic anti depressants and major tranquillisers, as well as the consumption of alcohol, may potentiate the BP lowering effects of MED2005; therefore, the PI must consider this carefully and include subjects at their discretion
3. Any presence of a symptomatic, active urinary tract infection diagnosed by the PI or their delegate at screening or during the study
4. Any presence of chronic indwelling urethral catheterisation or penile anatomical abnormalities (e.g. penile fibrosis) that would significantly impair EF
5. Any history of operations for Peyronie's disease
6. Primary hypoactive sexual desire or any history of hypogonadism
7. Any history of radical prostatectomy
8. Any history of severe/uncontrolled diabetes
9. Subjects taking two or more anti hypertensives for the treatment of BP
10. Hypersensitivity to GTN or to any of the excipients, or idiosyncratic reactions to other organic nitrates
11. Concomitant treatment with sildenafil citrate, tadalafil, vardenafil and other PDE 5 inhibitors
12. Subjects taking Alpha blockers
13. Subjects receiving testosterone pellets
14. Any penile surgery except circumcision
15. Any treatment with acetyl cysteine within 6 months
16. Any treatment with dihydroergotamine within 6 months
17. Postural hypotension, hypotension or uncorrected hypovolaemia, as the use of GTN in such states could produce severe hypotension or shock
18. Increased intracranial pressure (e.g. head trauma or cerebral haemorrhage) or inadequate cerebral circulation
19. Any history of migraine or recurrent headache
20. Aortic or mitral stenosis
21. Hypertrophic obstructive cardiomyopathy
22. Constrictive pericarditis or pericardial tamponade
23. Closed-angle glaucoma
24. Subjects with nursing partners, known pregnant partners or with partners who wish to become pregnant during the course of the study
25. Confirmed positive results from urine drug screen (amphetamines, benzodiazepines, cocaine, cannabinoids, opiates, barbiturates, tricyclic antidepressants and methadone) or from the alcohol breath test at screening (for clarification, any positive result from the urine drug screen or alcohol breath tests at screening will mean the subject will be excluded from the study). In the instance that a subject is using medication which may give a positive result, exclusion will be at the PI's discretion
26. Subject has recent (last 12 months) clinical evidence of alcoholism or drug abuse.
27. Subject has a positive screen for hepatitis B, consisting of hepatitis B surface antigen (HBsAG), hepatitis C antibody, and human immunodeficiency virus (HIV)
28. Any clinically significant abnormal laboratory, vital signs or other safety findings as determined by medical history, physical examination or other evaluations conducted at screening or on admission
29. Subjects unwilling to cease use of vacuum devices, intracavernosal injections, PDE-5s or other therapy for ED for the entire course of the study
30. Unwillingness of the subject or their partner to agree to make the required attempts at sexual intercourse during treatment period
31. Any history of unresponsiveness to PDE 5 treatment or significant side effects, excluding visual disturbances, with PDE 5s
32. Fewer than four attempts at sexual intercourse during the screening period
33. Subjects or their partners who are illiterate or are unable to understand the language in which the questionnaires are available
34. Subject has received any investigational product during the 90 days prior to dosing for this study
35. Subject or his partner cannot communicate reliably with the PI
36. Subjects with severe premature ejaculation (little or no control of ejaculation at the time of penetration)

Subjects are prohibited from participating in the open-label extension phase of the study if they meet any of the following exclusion criteria at the follow-up visit of the double-blind phase (Visit 6):

1. Subsequent to recruitment into the double-blind phase of the study, the development of any significant or serious cardiovascular, pulmonary, hepatic, renal, gastrointestinal, haematological, endocrinological, metabolic, neurological or psychiatric disease which, in the opinion of the PI, renders the subject unfit to continue in the open-label extension phase of the study
2. Subject using any medication that, in the opinion of the PI, is likely to affect the subject's ability to complete or participate in the open-label phase of the study.

   NB The concomitant medications listed as exclusion criteria for the study apply to the open-label extension phase. Certain concomitant medications; e.g. other vasodilators, calcium channel blockers, ACE inhibitors, beta blockers, diuretics, anti hypertensives, tricyclic anti depressants and major tranquillisers, as well as the consumption of alcohol, may potentiate the BP lowering effects of MED2005; therefore, the PI must consider this carefully and include subjects at their discretion
3. Any presence of a symptomatic, active urinary tract infection diagnosed by the PI or their delegate at the start of the open-label extension phase
4. Subsequent to recruitment into the double-blind phase of the study, the development of postural hypotension, hypotension or uncorrected hypovolaemia, increased intracranial pressure or inadequate cerebral circulation, any clinically significant vital signs or other safety findings as determined by medical history, physical examination or other evaluations conducted at Visit 6 prior to recruitment to the open-label phase

Ages: 18 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Male patients must have been in a heterosexual relationship with a female partner for a minimum of 6 months
Enrollment: 1005 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2019-07-21 (Actual); Study Completion 2020-01-17 (Actual)

PRIMARY OUTCOMES:
International Index for Erectile Function (IIEF) Questionnaire | Up to Week 64 of the study
  A questionnaire containing 15 questions divided into 5 domains; erectile function, orgasmic function, sexual desire, intercourse satisfaction, and overall satisfaction.
Sexual Encounter Profile (SEP) Questionnaire (Question 2) | Up to Week 64 of the study
  A questionnaire consisting of 5 items assessing the sexual events a patient experiences during sexual intercourse.
Sexual Encounter Profile (SEP) Questionnaire (Question 3) | Up to Week 64 of the study
  A questionnaire consisting of 5 items assessing the sexual events a patient experiences during sexual intercourse.

SECONDARY OUTCOMES:
Self-Esteem and Relationship (SEAR) Questionnaire | Up to Week 12 of the study.
  A questionnaire to support the validity and reliability for measuring sexual relationship satisfaction, satisfaction, confidence, and self-esteem in men with erectile dysfunction.
Global Assessment Questionnaire (GAQ) | Up to Week 12 of the study.
  A questionnaire that allows patients and their partners to rate (yes or no) an improvement in erectile function.
International Index for Erectile Function (IIEF) Questionnaire (additional domains) | Up to Week 64 weeks of the study.
  A questionnaire containing 15 questions divided into 5 domains; erectile function, orgasmic function, sexual desire, intercourse satisfaction, and overall satisfaction.
Sexual Encounter Profile (SEP) Questionnaire (Questions 1, 4 & 5) | Up to Week 64 of the study.
  A questionnaire consisting of 5 items assessing the sexual events a patient experiences during sexual intercourse.
Sexual Encounter Profile (SEP) Questionnaire | Up to Week 64 of the study
  A questionnaire consisting of 5 items assessing the sexual events a patient experiences during sexual intercourse.
Patient Global Impression of Severity (PGI-S) | Up to Week 12 of the study.
  A one item questionnaire to rate the severity of a patient's erectile dysfunction. This is a single-state 5-point categorical scale.
Patient Global Impression of Change (PGI-C) | Up to Week 12 of the study
  A one item questionnaire to rate a perceived change in a patient's erectile function. This is a transitional 7-point categorical scale.
Onset and duration of action (erection) and erection hardness | Up to Week 12 of the study
  A questionnaire asking both the patient and the patient's partner about the onset and duration of action of the patient's erection.
Usage and application | Up to Week 12 of the study
  A questionnaire has 5 items to assess the usage and application of the investigation product.

CONTACTS AND LOCATIONS:
Overall Officials: Tim J Holland, MBA, Study Director — Clinical Development Director
Locations (53):
- Bulgaria (5):
  - UMHAT Burgas EAD, Burgas
  - Multiprofile Hospital for Active Treatment, Pleven
  - University Multiprofile Hospital for Active Treatment, Plovdiv
  - Urology Office Diagnostic-Consultative Center, Varna
  - Medical Center Biomed, Vidin
- Czechia (3):
  - URAN MUDr.Jan Hiblbauer s.r.o, Hradec Králové
  - ANDROGEOS, spol. s.r.o., Prague
  - Urosante s.r.o., Prague
- Georgia (4):
  - LTD Gormedi, Gori
  - LTD Gidmedi, Tbilisi
  - LTD Multiprofile Clinic Consilium Medulla, Tbilisi
  - LTDHealth House, Tbilisi
- Hungary (4):
  - Synexus Magyarorszag Kft, Budapest
  - Civis Egeszseghaz, Debrecen
  - Korona Prevent-Med Kft., Sopron
  - Aranyklinika, Szeged
- Latvia (3):
  - Latgales Urology Center, Daugavpils
  - V. Lietuviesa Private Practice, Riga
  - Vidzemes Hospital, Valmiera
- Poland (4):
  - Indywidualna Specjalistyczna Praktyka Lekarska Dr Adam Sipinski, Katowice
  - PROVITA Specjalistyczna Praktyka Ginekologiczno-Seksuologiczna, Lublin
  - Indywidualna Specjalistyczna Praktyka Lekarska, Szczecin
  - Gabinet Lekarski Ryszard Smolinski, Wroclaw
- Russia (18):
  - Regional Budgetary Healthcare Institution "Ivanovskaya Regional Clinical Hospital", Ivanovo
  - CJSC "Nasledniki", Moscow
  - Federal State Budgetary Institution "National Medical Research Center of Obstetrics, Gynecology and Perinatology n.a. acad. V.I. Kulakov" of the Ministry of Healthcare of the Russian Federation, Moscow
  - FSBEI HE "Russian National Research Medical University n.a. N.I. Pirogov" of the Ministry of Healthcare of the Russian Federation, Russian Gerontological Scientific and Research Center, Moscow
  - LLC "Bessalar Clinic", Moscow
  - LLC "Unimed-S", Moscow
  - State Budgetary Institution "Hospital for War Veterans", Rostov-on-Don
  - Federal State Budgetary Educational Institution of Higher Education "North-Western State Medical University n.a. I.I. Mechnikov" of the Ministry of Healthcare of the Russian Federation, Saint Petersburg
  - LLC "Medical center PRIME ROSE", Saint Petersburg
  - LLC "Sanavita", Saint Petersburg
  - Llc <<Mart>>, Saint Petersburg
  - Medicosanitary Department No.70, branch of Saint-Petersburg State Unitary Institution of road passenger transport, Saint Petersburg
  - Research Center "Eco-Safety", Saint Petersburg
  - Saint Petersburg State Budgetary Healthcare Institution "City Polyclinic No. 4", Saint Petersburg
  - Clinical Hospital n.a. S.R. Mirotvortseva of the Federal State Budgetary Educational Institution of Higher Education "Saratovskiy State Medical University n.a. V.I. Razumovskiy" of the Ministry of Healthcare of the Russian Federation, Saratov
  - Federal State Budgetary Educational Institution of Higher Education " Voronezhskiy State Medical University n.a. N.N. Burdenko" of the Ministry of Healthcare of the Russian Federation on the clinical base of Budgetary Healthcare Institution of Voronezhsk, Voronezh
  - SBHI of Leningradskaya region "Vsevolozhskaya Clinical Interdistrict Hospital", Vsevolozhsk
  - FSBEI HPE "Yaroslavskiy State Medical University" of The Ministry of Healthcare of the Russian Federation with clinical base in State Autonomous Institution of Yaroslavskaya region "Clinical Hospital No.9", Yaroslavl
- Slovakia (4):
  - Urologicka ambulancia, Košice
  - Urologicka ambulancia Urobet s.r.o., Malacky
  - Urologicka ambulancia Uroexam s.r.o., Nitra
  - Privatna urologicka ambulancia s.r.o., Trenčín
- Ukraine (8):
  - Municipal Establishment "Cherkasy Regional Hospital of Cherkasy Regional Council", Urology department, Cherkasy
  - Regional Clinical Hospital, Polyclinic Department, Ivano-Frankivsk
  - Kyiv Clinical Hospital on Railway Transport #1 of the branch "Health Center" of the public joint stock company "Ukrainian Railway", consulting and diagnostic center, Kyiv
  - State Institution "Institute of urology of the National Academy of Medical Science of Ukraine", policlinic department, Kyiv
  - State Institution "Institute of urology of the National Academy of Medical Sciences of Ukraine", Department of Sexual Pathology and Andrology, Kyiv
  - "Ambulatory of General Practice-Family Medicine",LLC, Medical Center, Odesa
  - Private Small-Scale Enterprise Medical Centre "Pulse" , Therapeutic Department, Vinnytsia
  - Municipal Institution Central City Hospital №1 of Zhytomyr, consulting and medical department "Research center", Zhytomyr

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2018-07-27): https://cdn.clinicaltrials.gov/large-docs/92/NCT03813992/Prot_000.pdf